CLINICAL TRIAL: NCT04091373
Title: A Phase 1, Randomized, Open-label, Single Center, Three Period Cross-over Study to Evaluate the Pharmacokinetics of Single Dose Administration of Cotadutide in Healthy Subjects
Brief Title: A Study Investigating the Pharmacokinetics of a Single Dose Administration of Cotadutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D5670C00025
Record Dates: First submitted 2019-08-28; First posted 2019-09-16 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Sequence 1 (Experimental): 100ug SC injection cotadutide in the upper arm on Day 1, in the lower abdomen on Day 8, and in the thigh on Day 15
  Interventions: Combination Product: cotadutide multidose pen injection
- Sequence 2 (Experimental): 100ug SC injection cotadutide in the thigh on Day 1, in the upper arm on Day 8, and in the lower abdomen on Day 15
  Interventions: Combination Product: cotadutide multidose pen injection
- Sequence 3 (Experimental): 100ug SC injection cotadutide in the lower abdomen on Day 1, in the thigh on Day 8, and in the upper arm on Day 15
  Interventions: Combination Product: cotadutide multidose pen injection
- Sequence 4 (Experimental): 100ug SC injection cotadutide in the thigh on Day 1, in the lower abdomen on Day 8, and in the upper arm on Day 15
  Interventions: Combination Product: cotadutide multidose pen injection
- Sequence 5 (Experimental): 100ug SC injection cotadutide in the lower abdomen on Day 1, in the upper arm on Day 8, and in the thigh on Day 15
  Interventions: Combination Product: cotadutide multidose pen injection
- Sequence 6 (Experimental): 100ug SC injection cotadutide in the upper arm on Day 1, in the thigh on Day 8, and in the lower abdomen on Day 15
  Interventions: Combination Product: cotadutide multidose pen injection

INTERVENTIONS:
Combination Product: cotadutide multidose pen injection — SC injection in the upper arm
Combination Product: cotadutide multidose pen injection — SC injection in the lower abdomen
Combination Product: cotadutide multidose pen injection — SC injection in the thigh

SUMMARY:
This is a randomized, open label, cross-over study in healthy adult subjects to investigate cotadutide exposure after subcutaneous injection at 3 different anatomical sites. The study will be conducted at a single US center. Each subject will be randomized to receive a single SC dose of 100 μg cotadutide via a pen device according to 6 sequences of dosing. Each SC injection will be administered by a health care provider at a different injection site (arm, thigh, or abdomen) in each period. SC injection in the abdomen will be used as the reference treatment to determine the relative PK of cotadutide 100 μg SC injections in the arm and thigh. Each SC injection of cotadutide will be separated by 7 days washout. Blood samples for PK analyses of cotadutide will be taken pre dose and at 11 time points up to 48 hours after dosing (Days 3, 10, and 17).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 through 60 years (inclusive) at the time of screening.
2. Electronic and/or written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
3. BMI between 19 and 30 kg/m2 (inclusive) at screening.
4. Good general health as judged by the investigator, based on medical history, physical examination including 12 lead electrocardiogram (ECG), vital signs, and blood and urinary laboratory assessments.
5. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of investigational product, and must not be breastfeeding.
6. Female subjects of childbearing potential who are sexually active with a male partner must be using at least one highly effective method of contraception from screening and up to 4 weeks after the last dose of investigational product. As applicable, at least one method must be in effect prior to receiving the first dose of investigational product.

Exclusion Criteria:

1. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, put the subject at risk, influence the subject's ability to participate, or affect interpretation of subject safety or study results.
2. Inflammatory bowel disease, gastroparesis or other severe disease or surgery affecting the upper GI tract, which may affect gastric emptying or could affect the interpretation of safety and tolerability data.
3. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2; eGFR will be determined by the chronic kidney disease - epidemiology collaboration (CKD-EPI) equation.
4. BP and heart rate in supine position outside the ranges of 90 140 mmHg systolic, 50-90 mmHg diastolic and heart rate 40-100 beats/min following a 10 minute rest period.
5. Active hepatitis B, measured by positive tests of surface antigen HBsAg and/or active hepatitis C, measured by positive hepatitis C virus antibody tests.
6. Positive human immunodeficiency virus (HIV) antibodies.
7. Subjects with a history of acute or chronic pancreatitis.
8. Subjects with a history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, and subjects with a screening/baseline serum calcitonin ≥ 50 ng/L.
9. Signs or symptoms of severe hepatic impairment AND any of the following laboratory values at screening: Aspartate transaminase (AST) ≥ 3 × upper limit of normal (ULN), alanine transaminase (ALT) ≥ 3 × ULN, or total bilirubin (TBL) ≥ 2 × ULN. Alternatively, AST ≥ 5 × ULN, ALT ≥ 5 × ULN, or TBL ≥ 2 × ULN regardless of signs and symptoms. An isolated increase in TBL in subjects with known Gilbert's syndrome is not a reason for exclusion.
10. Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss), a history of type 1 diabetes mellitus or diabetic ketoacidosis.
11. History of neoplastic disease within 5 years prior to screening except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer.
12. Known or suspected allergy to cotadutide, any component of the formulation, or related products.
13. Use of any prescription or nonprescription medication, with the exception of permitted concomitant medications, within the last 72 hours prior to Day 1.
14. History of alcoholism or drug abuse during the last 12 months.
15. Current smoker of cigarettes or other tobacco products.
16. Habitual excessive consumption of methylxanthine containing (theophylline, caffeine, or theobromine) beverages and foods (eg, coffee, tea, red bull, cola, chocolate) as judged by the investigator.
17. Blood donation within the last 3 months.
18. Participation in any other study investigating other products or involving blood sampling within the past 30 days.
19. Potentially noncompliant or uncooperative, as judged by the investigator.
20. Substance dependence likely to impact subject safety or compliance with study procedures, to include a positive test result for drugs of abuse and/or alcohol at screening or prior to administration of investigational product on Day 1.
21. Psychiatric illness such that subjects have been committed to an institution by way of official or judicial order.
22. Involvement of any AstraZeneca, MedImmune, the contract research organization, or the study center employee or their close relatives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve | 48 hours
  To evaluate exposure following a single subcutaneous dose of cotadutide at each of 3 different sites of injection.

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration | 48 hours
  To evaluate exposure following a single subcutaneous dose of cotadutide at each of 3 different sites of injection.
Area under the plasma concentration time curve from zero to infinity | 48 hours
  To evaluate exposure following a single subcutaneous dose of cotadutide at each of 3 different sites of injection
Time to maximum observed plasma drug concentration | 48 hours
  To evaluate exposure following a single subcutaneous dose of cotadutide at each of 3 different sites of injection
Terminal phase elimination half life | 48 hours
  To evaluate exposure following a single subcutaneous dose of cotadutide at each of 3 different sites of injection
Apparent clearance | 48 hours
  To evaluate exposure following a single subcutaneous dose of cotadutide at each of 3 different sites of injection.
Anti drug antibody incidence and titer | 43 Days
  To evaluate the immunogenicity of a single subcutaneous dose of cotadutide at each of 3 different sites of injection
Incidence of treatment-emergent adverse events, including those related to changes in vital signs (including body temperature, heart rate, blood pressure) and safety laboratory evaluations (including hematology, chemistry, plasma glucose, urinalysis). | 43 Days
  To evaluate the safety and tolerability of a single subcutaneous dose of cotadutide at each of 3 different sites of injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home